CLINICAL TRIAL: NCT04418453
Title: Rural Expansion of Medication Treatment for Opioid Use Disorder (Rural MOUD): Phase 1 Feasibility Study (CTN-0102)
Brief Title: Rural MOUD Telemedicine in Primary Care Phase 1
Acronym: Feasibility
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Yih-Ing Hser, Principal Investigator, University of California, Los Angeles
Other Study IDs: RMOUD1; 1UG1DA049435 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-06-05 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Opioid-use Disorder
Keywords: Medication treatment for opioid use disorder; Telemedicine; Rural areas
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Primary Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Integration of telemedicine in primary care settings for MOUD: Primary care providers may refer OUD patients to receive telemedicine for MOUD
  Interventions: Other: Integration of telemedicine for MOUD in primary care

INTERVENTIONS:
Other: Integration of telemedicine for MOUD in primary care — Patients with opioid use disorder in rural primary care settings may be referred to receive telemedicine for medication treatment for opioid use disorder

SUMMARY:
The feasibility study (Phase 1) will examine the implementation of telemedicine (TM) in six rural clinics in two states/regions with varying levels of OBOT capacity.

DETAILED DESCRIPTION:
The dramatic increases in opioid overdose deaths across the nation, particularly in rural areas, call for a rapid expansion of access to medication treatment for opioid use disorder (MOUD).There is a need to study effective ways to expand treatment access and improve retention on MOUD in rural areas highly impacted by OUD. Telemedicine (TM) for MOUD offers an alternative or supplementary approach to delivering MOUD that may be suitable for rural clinics and patients with OUD.

The objectives of the feasibility study are to study ways of incorporating TM into primary care clinics and to evaluate the associated outcomes, based on EHRs from the clinics and the TM vendor (i.e., patient days on MOUD) and participant surveys (e.g., opioid use). Additional outcomes of the feasibility study are feasibility and acceptability assessed from the perspectives of providers and participants via focus groups. A patient registry will be established in each clinic to track patients with OUD diagnoses, and those in the registry will be provided the opportunity to consent for sharing identified EHRs and participating in the follow-up surveys.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years old, inclusive, at the time of the qualifying visit
* with OUD diagnosis
* At least 1 visit to the participating clinics from 9 months before and 6 months after the date of intervention implementation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients
Sampling Method: Non-Probability Sample
Enrollment: 36762 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Patient days on MOUD from Electronic Health Records (EHR) | 9 months
  Number of days patients receive MOUD based on EHR data

SECONDARY OUTCOMES:
Number of OUD patients initiating/receiving MOUD | 9 months
  Number of OUD patients initiating/receiving MOUD

OTHER OUTCOMES:
Treatment retention | 3 months
  Number of patients retained in treatment at 3 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Ing Hser, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (7):
- United States (7):
  - St. Mary's Hospital and Clinics, Cottonwood, Idaho
  - Syringa Hospital and Clinics, Grangeville, Idaho
  - Penobscot Community Health Care, Belfast, Maine
  - Hometown Health Center, Dexter, Maine
  - Penobscot Community Health Care, Winterport, Maine
  - Providence Northeast Washington Medical Group, Colville, Washington
  - Ferry County Health, Republic, Washington

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant survey data will be shared on the NIDA Data Share website.
Access Criteria: The data on NIDA Data Share website are accessible to anyone.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Background] Hser YI, Mooney LJ, Baldwin LM, Ober A, Marsch LA, Sherman S, Matthews A, Clingan S, Fei Z, Zhu Y, Dopp A, Curtis ME, Osterhage KP, Hichborn EG, Lin C, Black M, Calhoun S, Holtzer CC, Nesin N, Bouchard D, Ledgerwood M, Gehring MA, Liu Y, Ha NA, Murphy SM, Hanano M, Saxon AJ. Care coordination between rural primary care and telemedicine to expand medication treatment for opioid use disorder: Results from a single-arm, multisite feasibility study. J Rural Health. 2023 Sep;39(4):780-788. doi: 10.1111/jrh.12760. Epub 2023 Apr 19. PMID 37074350
- [Derived] Flores JM, Kan E, Mooney LJ, Pham H, Zhu Y, Wolitzky-Taylor K, Hser YI. Medications for Opioid Use Disorder Among Transition Age Youth Compared to Adults 26 or Older in Rural Settings. JAACAP Open. 2024 Feb 28;2(4):231-238. doi: 10.1016/j.jaacop.2024.02.001. eCollection 2024 Dec. PMID 39697397
- [Derived] Pham H, Ober A, Baldwin LM, Mooney LJ, Zhu Y, Fei Z, Hser YI. Social Determinants of Health and Continuity of Medications for Opioid Use Disorder Among Patients Receiving Treatment in Rural Primary Care Settings. J Addict Med. 2024 May-Jun 01;18(3):331-334. doi: 10.1097/ADM.0000000000001274. Epub 2024 Feb 5. PMID 38315721
- [Derived] Osterhage KP, Hser YI, Mooney LJ, Sherman S, Saxon AJ, Ledgerwood M, Holtzer CC, Gehring MA, Clingan SE, Curtis ME, Baldwin LM. Identifying patients with opioid use disorder using International Classification of Diseases (ICD) codes: Challenges and opportunities. Addiction. 2024 Jan;119(1):160-168. doi: 10.1111/add.16338. Epub 2023 Sep 15. PMID 37715369